CLINICAL TRIAL: NCT05733884
Title: Soft Peripheral Contact Lens for Eye Elongation Control (SPACE):1-year Results of a Double-blinded Randomized Con-trolled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS1-20136
Record Dates: First submitted 2023-01-16; First posted 2023-02-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Soft Contact Lens
Keywords: axial length; children; myopia control; soft contact lens; clinical trials
MeSH Terms: interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Disposable Multifocal Soft Contact lenses, PEGAVISION, Taiwan (Experimental): Subjects will be asked to wear the lenses for 8 hours a day, at least 7 days a week. Contact lenses are worn and replaced every day. All subjects will be followed for 1 year after device allocation and will undergo brief clinical assessments at 1 day, 1 week, 1, 3, 6, 9, and 12 months.
  Interventions: Other: soft contact lens
- Omafilcon A, dual-focus optical design, USA (Active Comparator): Subjects will be asked to wear the lenses for 8 hours a day, at least 7 days a week. Contact lenses are worn and replaced every day. All subjects will be followed for 1 year after device allocation and will undergo brief clinical assessments at 1 day, 1 week, 1, 3, 6, 9, and 12 months.
  Interventions: Other: soft contact lens

INTERVENTIONS:
Other: soft contact lens — soft contact lens

SUMMARY:
A prospective, randomised, double-blinded clinical trial was conducted including 115 children (55 male and 60 female) aged 8 to 15 years. The newest multifocal contact lenses were assigned to experimental group, and another commercial dual-focus optical designed contact lenses were assigned to control group to be worn for at least 8 hours per day, 7 days a week, for a period of 1 year. All contact lenses were replaced with new lenses every day. Measurements obtained using a LogMAR vision meter, including automated computerised optometry, handheld retinoscopy, high (96%) and low (12%) contrast sensitivity visual acuity values at a distance, and near-visible acuity values were used to evaluate the corneal curvature using a corneal mapper. Additionally, the axial length(AXL) of the eye was measured, and the tear quality was assessed using a slit lamp, including tear break-up time, tear river height, and observation of blink frequency. Furthermore, the eye's anterior surface was examined by slit lamp using the Efron grading scale.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 8 and 15 (both 8 and 15 years old).
* Subject's best corrected visual acuity must be at least LogMAR 0.10 or higher in both eyes.
* The subject's eyes must be healthy and normal, and "normal eyes" is defined as having the following characteristics.

  1. Based on the slit-lamp examination results of the screening clinic, determined that the infection of the conjunctiva, eyelids and accessory organs was less than Grade 2 (mild).
  2. No structural abnormality of the eyelid, conjunctiva or accessory organ tissue.
  3. Slit lamp findings must be less than Grade 1 (mild) and the cornea must not show: edema, staining, clouding, or vascularization according to the slit lamp findings of the screening clinic.
  4. No iritis.
  5. There are no other active eye diseases that are not suitable for contact lens wear.
* No topical eye drops are currently being used.
* The subject and his/her legal representative (if the subject is under 20 years old) are willing to sign the subject's consent form.
* Legal guardians of subjects under 12 years of age are willing to sign the informed consent form.
* Meet the following refractive criteria determined by cycloplegic autorefraction at baseline

  1. Spherical equivalent refractive error: between -0.75 and -6.00 D inclusive
  2. Astigmatism: ≤-0.75 D
  3. Anisometropia: <1.00 D

Exclusion criteria:

* Participants with certain eye diseases that may affect their eye health or may be aggravated by the test product.
* Those who are unable to comply with regular tracking and inspection.
* Subject is currently participating, or has participated in another drug trial within 4 weeks prior to enrollment in this trial.
* Subject has undergone any eye surgery or corneal surgery.
* Subject has used systemic steroids, other systemic medications that may significantly affect vision or recovery, ophthalmic steroids, eye ointments, or pupil dilators (except for examination pupil dilators) within 2 weeks prior to trial entry.
* Those who are unable to cooperate with regular tracking and inspection.
* Participants with poor hygiene practices that may compromise safety during the trial or be inconsistent with the participant's best interests.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Spherical Equivalent Refraction (SER) | 12 months
  The change in spherical equivalent refraction (SER) measured by cycloplegic autorefraction over 12 months.

SECONDARY OUTCOMES:
Axial Eye Length (AXL) | 12 months
  The change in axial eye length (AXL) measured over 12 months. Axial length is measured after cycloplegia using optical biometry.

OTHER OUTCOMES:
Primary safety Endpoints | 12 months
  All dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=severe findings. Epithelial edema, epithelial microcysts, corneal staining, limbal & bulbar injection, conjunctival abnormalities, corneal neovascularization and infiltrates will be measured.(700GL Slit Lamp, Takagi Europe)

CONTACTS AND LOCATIONS:
Overall Officials: Min yen Hsu, PhD, Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No